CLINICAL TRIAL: NCT03656458
Title: Effects of Balance Training on Fall Risk and Mobility in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Furqan Ahmed Siddiqi, Associate Dean (Academics) FUIRS, Foundation University Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUI/CTR/2018/1
Record Dates: First submitted 2018-08-13; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Fall
Keywords: Impaired Balance; Geriatrics; Balance Training; Dynamic Stability Training; Fall Risk; Berg Balance Scale; Physical Therapy; Forward Reach Test
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was not aware regarding the allocation of participants to study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group A (Active Comparator): Warm Up followed by Conventional Balance Training (Internal and External Perturbations)
  Interventions: Other: Warm Up; Other: Conventional Balance Training
- Control Group B (No Intervention): Control group. No intervention given to participants.
- Experimental Group (Experimental): Warm Up followed by Biodex Balance Training
  Interventions: Other: Warm Up; Other: Biodex Balance Training

INTERVENTIONS:
Other: Warm Up — 10 low jumps 5 Illiopoase Stretches 5 L/L Abductor Stretches 10 Trunk rotations 10 Should Circumduction Clock wise/Counter clockwise 10 Cervical Rotations Clockwise/Counter Clockwise
  Arms: Control Group A; Experimental Group
Other: Conventional Balance Training — Internal Protuberances:
  1. Looking up/Looking down/looking over the shoulder (Rt. /Lt.) 10 Reps Each
  2. Looking behind over the shoulder (Rt. /Lt.)10 Reps
  3. Looking Up with overhead Upper Limb Flexion. 5 Reps
  4. Reaching out of Base of support (Rt. /Lt. / midline Cross) 10 Reps Each
  5. Side to Side weight Shifting 10 Reps
  6. Standing on toes/Heels 10 Reps each
  External Protuberance:
  1. Tuck forward/ Backward/ Sideways(Rt. /Lt.) 10 reps Each
  2. Bosu Ball Training
  Arms: Control Group A
Other: Biodex Balance Training — Biodex Balance Training Using Biodex Balance System SD
  Arms: Experimental Group

SUMMARY:
Pakistan is a country devoid of health-care facilities and training programs on fall prevention. There is lack of research, awareness and implication of geriatric rehabilitation on elderly population addressing balance and fall risk assessment however very few cross-sectional studies of poor quality evidence are available on this issue. To best of investigators' knowledge, no interventional studies have been conducted in our country so far on this topic. . We aim to use a integrated method of balance training that uses patients judgment, visual feedback, proprioception and balance training with the help of new technology/devices to improve balance. And compare it to conventional treatment. We also aim to assess risk factors of fall in geriatric population, decreasing risks of falls and increasing awareness regarding geriatric rehabilitation and balance training.

DETAILED DESCRIPTION:
Balance is use of multiple systems of the body including auditory, motor, visual, vestibular and nervous to keep body staying inside limits of stability. It includes maintaining posture under different conditions in standing or sitting, ability to facilitate movement and to recover and stay in limits of stability after external (Trip, push, slip) and internal (body movements) protuberance. Impaired balancing system of body results in increased risk of fall which is major cause of mortality and morbidity in geriatric population.

A report of 2014 stated that Pakistan has 12.13 million population of Age 60 years and above which is expected to rise to 17.53 Million by year 2025. According to a study 30-50 % of population of age 65 years and above have some problems with balance. Another study states that 75 % of people aging 70 years and above have balance impairments which leads to fall. Additionally number of conditions including poly pharmacy, female gender, visual problems, environmental problems and cognitive issue contribute to in fall risk and balance problems. One of the major goal of Balance re-education is to decrease fall risk. Literature has suggested that one of the most effective methods of reducing falls in geriatric population is to prophylactically intervene on multiple risks factors of fall. This includes outpatient balance training and fall risk assessment.

Force plate systems and mirrors which are the part of visual biofeedback are often used for treatment of balance disorders but are found to have no difference in educating compared to conventional management. In current era technology has advances to a great extend and new systems that quantifies balance and provide a reliable and valid data regarding balance which then can be used in formation of balance training plan. These systems can also be used for treatment purposes and also have various visual feedback systems for more educational benefits. One of these systems is Biodex balance system which is used for balance and postural reduction, increase proprioception, somatosensory and neuromuscular control. It incorporates patient data saving and printing system for record management and uses an integrated system which involves patient in activities of re-education with relation to visual feedback to accommodate body accordingly.

As mentioned earlier Falls result in high morbidity and mortality among geriatric population which leads to increased costs and need for rehabilitation services. Falls are brought about by detrimental effects of aging on postural control as a result of deterioration in neuromuscular and sensory mechanisms, physical inactivity, pre-existing pathology and use of medications. However, balance training and exercise interventions tend to decrease risk of falling and eventually fall itself. Moreover, conventional balance training programs have decreased adherence; hence, sensor-based training programs have been advocated. These programs have quiet good advantages including visual feedback with interactive environment and targeted interventions. This exercise system incorporates human-computer interface providing a three-dimensional and real-time feedback.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of age 60 -80 years
* Both male and females

Exclusion Criteria:

* Musculoskeletal conditions

  * Fractures
  * Severe arthritis
* Neurological conditions

  * Epilepsy
  * Parkinson
  * Alzheimer's disease
  * Impaired cognition
* Other systemic diseases or co-morbidities

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Berg balance scale - Change is being assessed | Pre-treatment (Base line), First Follow Up (2 weeks), Second Follow Up (4 weeks), Third Follow Up (6 weeks) and at Final Follow Up (8 weeks)
Quantitative measure of balance via Biodex balance system - Change is being assessed | Pre-treatment (Base line), First Follow Up (2 weeks), Second Follow Up (4 weeks), Third Follow Up (6 weeks) and at Final Follow Up (8 weeks)
Forward reach test - Change is being assessed | Pre-treatment (Base line), First Follow Up (2 weeks), Second Follow Up (4 weeks), Third Follow Up (6 weeks) and at Final Follow Up (8 weeks)
Timed Up and Go Test - Change is being assessed | Pre-treatment (Base line), First Follow Up (2 weeks), Second Follow Up (4 weeks), Third Follow Up (6 weeks) and at Final Follow Up (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Furqan Ahmed Siddiqi, BSPT, PP-DPT, PhD, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancini M, Horak FB. The relevance of clinical balance assessment tools to differentiate balance deficits. Eur J Phys Rehabil Med. 2010 Jun;46(2):239-48. PMID 20485226
- [Background] Sibley KM, Straus SE, Inness EL, Salbach NM, Jaglal SB. Balance assessment practices and use of standardized balance measures among Ontario physical therapists. Phys Ther. 2011 Nov;91(11):1583-91. doi: 10.2522/ptj.20110063. Epub 2011 Aug 25. PMID 21868613
- [Background] Ambrose AF, Paul G, Hausdorff JM. Risk factors for falls among older adults: a review of the literature. Maturitas. 2013 May;75(1):51-61. doi: 10.1016/j.maturitas.2013.02.009. Epub 2013 Mar 22. PMID 23523272
- [Background] Tinetti ME, Kumar C. The patient who falls: "It's always a trade-off". JAMA. 2010 Jan 20;303(3):258-66. doi: 10.1001/jama.2009.2024. PMID 20085954
- [Background] Geiger RA, Allen JB, O'Keefe J, Hicks RR. Balance and mobility following stroke: effects of physical therapy interventions with and without biofeedback/forceplate training. Phys Ther. 2001 Apr;81(4):995-1005. PMID 11276182
- [Background] Schoene D, Valenzuela T, Lord SR, de Bruin ED. The effect of interactive cognitive-motor training in reducing fall risk in older people: a systematic review. BMC Geriatr. 2014 Sep 20;14:107. doi: 10.1186/1471-2318-14-107. PMID 25240384
- [Background] Schwenk M, Grewal GS, Honarvar B, Schwenk S, Mohler J, Khalsa DS, Najafi B. Interactive balance training integrating sensor-based visual feedback of movement performance: a pilot study in older adults. J Neuroeng Rehabil. 2014 Dec 13;11:164. doi: 10.1186/1743-0003-11-164. PMID 25496052